CLINICAL TRIAL: NCT00469326
Title: Atorvastatin Pre-Treatment Influences the Risk of Percutaneous Coronary Intervention Study
Acronym: TIPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: University Hospital Motol, University Hospital Motol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KC EK-361/05
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; percutaneous coronary intervention; atorvastatin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- atorvastatin (Active Comparator): atorvastatin pre-treatment group (80mg atorvastatin two days before PCI)
  Interventions: Drug: Atorvastatin
- control (No Intervention): PCI without atorvastatin pretreatment
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — two days 80mg atorvastatin pre-treatment before PCI
  Other Names: Torvacard

SUMMARY:
This study investigates potential protective effect of atorvastatin pre-treatment in patient with stable coronary artery disease undergoing percutaneous coronary intervention (PCI). Patient are randomized to two groups: atorvastatin pre-treatment group (80mg atorvastatin two days before PCI) and control group (PCI without atorvastatin pretreatment). Endpoint is myocardial infarction measured by troponin I and creatine kinase myocardial band.

DETAILED DESCRIPTION:
Randomized studies have shown that pre-treatment with atorvastatin may reduced periprocedural myocardial in patient with stable angina during elective PCI. These data provide evidence-based support for using atorvastatin 7 days before PCI (dosage 40mg/d), alternatively three or more days (unknown dosage). We want to confirm this results for shorter pre-treatment period (two days) with dosage 80mg per day.

ELIGIBILITY:
Inclusion Criteria:

* stable angina in last month
* indication for percutaneous coronary intervention
* informed consent

Exclusion Criteria:

* acute coronary syndrome in last 14 days
* renal insufficiency (creatinine more 150 µmol/l)
* diseases severely limiting prognosis
* immunosuppressive treatment
* statin one month before randomization
* occlusion of the coronary artery
* previous participation in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
periprocedural myocardial infarction measured by troponin I level | 24 hours

SECONDARY OUTCOMES:
periprocedural myocardial infarction measured by creatine kinase myocardial band | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Josef Veselka, Prof., PhD., Study Chair — Department of Cardiology, Cardiovascular Center, University Hospital Motol, Prague, Czech Republic
Locations (1):
- Department of Cardiology, CardioVascular Center, University Hospital Motol, Prague, Czechia

REFERENCES:
- [Background] Pasceri V, Patti G, Nusca A, Pristipino C, Richichi G, Di Sciascio G; ARMYDA Investigators. Randomized trial of atorvastatin for reduction of myocardial damage during coronary intervention: results from the ARMYDA (Atorvastatin for Reduction of MYocardial Damage during Angioplasty) study. Circulation. 2004 Aug 10;110(6):674-8. doi: 10.1161/01.CIR.0000137828.06205.87. Epub 2004 Jul 26. PMID 15277322
- [Background] Briguori C, Colombo A, Airoldi F, Violante A, Focaccio A, Balestrieri P, Paolo Elia P, Golia B, Lepore S, Riviezzo G, Scarpato P, Librera M, Bonizzoni E, Ricciardelli B. Statin administration before percutaneous coronary intervention: impact on periprocedural myocardial infarction. Eur Heart J. 2004 Oct;25(20):1822-8. doi: 10.1016/j.ehj.2004.07.017. PMID 15474697
- [Derived] Veselka J, Zemanek D, Hajek P, Maly M, Adlova R, Martinkovicova L, Tomasov P, Tesar D. Effect of two-day atorvastatin pretreatment on long-term outcome of patients with stable angina pectoris undergoing elective percutaneous coronary intervention. Am J Cardiol. 2011 May 1;107(9):1295-9. doi: 10.1016/j.amjcard.2010.12.040. Epub 2011 Feb 23. PMID 21349484
- [Derived] Veselka J, Zemanek D, Hajek P, Maly M, Adlova R, Martinkovicova L, Tesar D. Effect of two-day atorvastatin pretreatment on the incidence of periprocedural myocardial infarction following elective percutaneous coronary intervention: a single-center, prospective, and randomized study. Am J Cardiol. 2009 Sep 1;104(5):630-3. doi: 10.1016/j.amjcard.2009.04.048. Epub 2009 Jun 24. PMID 19699335